CLINICAL TRIAL: NCT04564872
Title: A Multicenter, Randomized, Double-Blind, Active-Controlled Trial of the Efficacy and Safety of Adding HSK7653 to Metformin in Chinese Patients With Type 2 Diabetes and Inadequate Glycaemic Control
Brief Title: HSK7653 Metformin Add-on Study in Patients With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sichuan Haisco Pharmaceutical Group Co., Ltd (Industry)
Responsible Party: Sponsor
Organization: Haisco Pharmaceutical Group Co., Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HSK7653-302; CTR20201724 (Other: www.chinadrugtrials.org.cn)
Record Dates: First submitted 2020-09-14; First posted 2020-09-25 (Actual); Last update posted 2022-12-12 (Actual); Status verified 2022-12

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Linagliptin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- HSK7653 10 mg (Experimental)
  Interventions: Drug: HSK7653 10 mg Q2W
- HSK7653 25 mg (Experimental)
  Interventions: Drug: HSK7653 25 mg Q2W
- Linagliptin 5 mg (Active Comparator)
  Interventions: Drug: Linagliptin 5 mg QD

INTERVENTIONS:
Drug: HSK7653 10 mg Q2W — HSK7653 5 mg (2 tablets) and placebo 25 mg (1 tablet) Q2W, placebo of linagliptin 5 mg QD, oral, week 1 to week 24; HSK7653 25 mg Q2W, oral, week 25 to week 52.
  Arms: HSK7653 10 mg
Drug: HSK7653 25 mg Q2W — HSK7653 25 mg (1 tablet) and placebo 5 mg (2 tablets) Q2W, placebo of linagliptin 5 mg QD, oral, week 1 to week 24; HSK7653 25 mg (1 tablet) Q2W, oral, week 25 to week 52.
  Arms: HSK7653 25 mg
Drug: Linagliptin 5 mg QD — Linagliptin 5 mg QD, placebo of HSK7653 25 mg (1 tablet) and 5 mg (2 tablets) Q2W, oral, week 1 to week 24; HSK7653 25 mg Q2W, oral, week 25 to week 52.
  Arms: Linagliptin 5 mg

SUMMARY:
The purpose of this study is to assess the efficacy of HSK7653 (as an add-on to metformin) compared with linagliptin after 24 weeks, and the safety (up to 52 weeks) of HSK7653 in Chinese patients with Type 2 Diabetes who have inadequate glycemic control on diet/exercise therapy and metformin agent monotherapy.

DETAILED DESCRIPTION:
The treatment period is composed of a 24-week double-blind period (week 1-24) and a 28-week open-label period (week 25-52). During the double-blind period, participants will receive 10 mg or 25 mg dose of HSK7653, or linagliptin, and with matching placebo respectively. During the open-label period, all participants will receive 25 mg dose of HSK7653. All participants will receive a stable dose of metformin therapy in both the double-blind period and the open-label period.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 and ≤ 75 years, Male and female patients;
* Type 2 diabetes mellitus;
* Insufficient glycaemic control with diet/exercise therapy and metformin agent monotherapy;
* Did not receive regular long-term medication of oral hypoglycemic drugs (except metformin) or insulin within 1 year prior to informed consent;
* HbA1c in the range of ≥7.5 to ≤11.0% at screening;
* FPG < 15 mmol/L at screening;
* BMI (Body Mass Index) in the range of ≥ 18.0 kg/m² to ≤ 35.0 kg/m² at screening.

Exclusion Criteria:

* Diabetic ketoacidosis, hyperglycemia hypertonic state, serious complications of diabetes, myocardial infarction, stroke within 6 months prior to informed consent;
* History of severe endocrine disease, uncured cancer, acute pancreatitis prior to informed consent;
* Current hemoglobinopathy, uncontrolled hypertension, serious nephropathy or hepatopathy prior to informed consent;
* Serious gastrointestinal disease within 2 weeks prior to informed consent;
* Serious infection, trauma, and surgery within 3 months prior to informed consent;
* History of treatment with Dipeptidyl-Peptidase 4 (DPP-4) inhibitor, Glucose-dependent insulinotropic polypeptide (GIP) or Glucagon-like peptide-1 (GLP-1) receptor agonist;
* Treatment with drugs that affect glucose metabolism within 8 weeks prior to informed consent;
* Hemoglobin (HGB) < 10.0 g/dL(100 g/L);
* Alcohol abuse within 6 months or drug abuse history within 5 years prior to informed consent;
* Active infectious diseases;
* Participation in another trial with an investigational drug or instrument within 3 months prior to informed consent;
* Women who are nursing or pregnant, or subjects who have planned parenthood;
* Contraindication for empagliflozin or linagliptin;
* Other protocol-defined inclusion/exclusion criteria.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 465 (Actual)
Dates: Start 2020-11-13 (Actual); Primary Completion 2022-01-21 (Actual); Study Completion 2022-08-29 (Actual)

PRIMARY OUTCOMES:
HbA1c Change From Baseline at Week 24 | Baseline and week 24
  Change From Baseline in Hemoglobin A1c (HbA1c) at Week 24

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | Baseline, week 24 and week 52
  The incidence of Treatment-Emergent Adverse Events over time (at week 24 and week 52)
Percentage of Patients With HbA1c <7.0% | Baseline, week 24 and week 52
Percentage of Patients With HbA1c <6.5% | Baseline, week 24 and week 52
FPG Change From Baseline at Week 24 and Week 52 | Baseline , week 24 and week 52
2h-PPG Change From Baseline at Week 24 and Week 52 | Baseline, week 24 and week 52
Weight Change From Baseline at Week 24 and Week 52 | Baseline, week 24 and week 52
Fasting C-peptide Change From Baseline at Week 24 and Week 52 | Baseline, week 24 and week 52
Insulin Sensitivity Change (Calculated by HOMA-IS) From Baseline at Week 24 and Week 52 | Baseline, week 24 and week 52
Pancreatic β-cell function Change (Calculated by HOMA-β) From Baseline at Week 24 and Week 52 | Baseline, week 24 and week 52
Percentage of Patients Required Use of Rescue Therapy or Dropout due to Hyperglycemia and Week 52 | Baseline, week 24 and week 52

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Inner Mongolia Baogang Hospital, Baotou, Inner Mongolia

IPD SHARING:
Plan to Share IPD: No